CLINICAL TRIAL: NCT04339309
Title: Comparison Between Two Non-surgical Periodontal Treatment Procedures With and Without Interdental Hygiene Devices in Periodontitis Patients: a Longitudinal Prospective Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Karim Fawzy El-Sayed, Assistant Professor of Periodontology, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDB Kiel-Cairo15
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kiel Center (Active Comparator): Non-surgical periodontal treatment with interdental hygiene devices in periodontitis patients.
  Interventions: Procedure: Non-surgical periodontal treatment with interdental hygiene devices
- Cairo Center (Active Comparator): Non-surgical periodontal treatment without interdental hygiene devices in periodontitis patients.
  Interventions: Procedure: Non-surgical periodontal treatment without interdental hygiene devices

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment with interdental hygiene devices
  Arms: Kiel Center
Procedure: Non-surgical periodontal treatment without interdental hygiene devices
  Arms: Cairo Center

SUMMARY:
Periodontitis is treated by regularly clearance of the disease-causing biofilm through domestic care and dental measures (Petersilka et al., 2002, Herrera et al., 2008). Healthy gums have intact papillae occluding the interdental area. Successful brushing cleans these areas; the prophylaxis of gingivitis for such patients does therefore not require special aids. In contrast, initial attachment loss as a result of inflammation or restorative therapy leads to additional cleaning needs, since the normal brush is not able to clean interdental areas as successful as vestibular and oral surfaces (Dörfer and Staehle, 2010).

It can be said that interdental brushes are the most effective tools for cleaning interdental spaces (Salzer et al., 2015). Compared with a toothbrush, they are the only tool showing better results of plaque removal and reduction of gingivitis (Slot et al., 2008). Therefore their use should not be restricted to older people with already reduced interdental papillae. A big advantage is that interdental brushes are generally easy to use. If brush sizes are chosen correctly, insertion and multiple forward and backward movement is sufficient to obtain com- plete cleaning of the interproximal surfaces. Additional cleaning by other means such as dental floss is not always necessary because interdental brushes clean approximal and subgingival surfaces sufficiently, providing the size was chosen correctly (Dörfer and Staehle, 2010).

Due to the above mentioned coherences and associations, this study includes the hypothesis that patients with periodontitis would benefit from the instruction and motivation of interdental brushes within the active periodontitis therapy in comparison to a periodontitis therapy without the instructed domestic interdental hygiene by a stronger reduction of clinical inflammatory characteristics (Salzer et al., 2015). The corresponding Zero-Hypothesis says that no difference would be found between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Generalized chronic periodontitis (CP)
* Generalized aggressive periodontitis (AgP)
* Availability for non-surgical periodontal therapy and reevaluation after 3±1 months.
* Moderate to advanced severity of periodontitis (≥30% of the sites with attachment loss ≥3mm)
* Age: 18 - 70 years
* ≥16 scorable teeth, without root caries

Exclusion Criteria:

* Localized chronic or aggressive periodontitis (<30% diseased teeth of all teeth)
* Smoking
* Tumour(s) of the soft or hard tissues of the oral cavity.
* Systematic disease, which include specific conditions to treat (e.g. prophylaxis of endocarditic)
* Women who are aware of being pregnant or who are breastfeeding.
* Forms of acute necrotizing ulcerating periodontitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 3 months
  Bleeding on probing (BOP) will be measured at least after the measurement of the CAL through recording bleeding sign at the site of clinical probing (six sites of each teeth).

SECONDARY OUTCOMES:
Probing pocket depth | 3 months
  Probing Pocket Depth (PPD) at every site will be assessed as the distance (mm) from the gingival margin to the apical end of the pocket using a PCP UNC-15 probe (Hu-Friedy, Chicago Ill, USA). The probe will be inserted parallel to the root surface and directed apically toward the perceived location of the apex of the root until slight resistance is felt. Probe recordings will be rounded off to the nearest millimeter mark. PPDs are measured at six areas of the tooth. These are the disto-vestibular, vestibular, mesio-vestibular, disto-lingual, lingual and the mesio-lingual. First the vestibular surface is probed and scored. Thereafter, the lingual surface is probed and scored.
Clinical attachment level (CAL) | 3 months
  The CAL at every site will be measured as the distance between the cemento-enamel junction (CEJ) and the apical end of the pocket using a PCP UNC-15 probe (Hu-Friedy, Chicago Ill, USA). The probe will be placed parallel to the tooth surface and probe recordings will be rounded off to the nearest millimeter mark. A score is given to six areas of the tooth. These are the disto-vestibular, vestibular, mesio-vestibular, disto-lingual, lingual and the mesio-lingual. First the vestibular surface is probed and scored. Thereafter, the lingual surface is probed and scored.
Antibiotic use | 3 months
  Measure whether antibiotics are used or not during the treatment phase by a questionnaire

REFERENCES:
- [Background] Behle JH, Papapanou PN. Periodontal infections and atherosclerotic vascular disease: an update. Int Dent J. 2006 Aug;56(4 Suppl 1):256-62. doi: 10.1111/j.1875-595x.2006.tb00110.x. PMID 16972401
- [Background] Herrera D, Alonso B, Leon R, Roldan S, Sanz M. Antimicrobial therapy in periodontitis: the use of systemic antimicrobials against the subgingival biofilm. J Clin Periodontol. 2008 Sep;35(8 Suppl):45-66. doi: 10.1111/j.1600-051X.2008.01260.x. PMID 18724841
- [Background] Jared H, Zhong Y, Rowe M, Ebisutani K, Tanaka T, Takase N. Clinical trial of a novel interdental brush cleaning system. J Clin Dent. 2005;16(2):47-52. PMID 16170976
- [Background] Petersilka GJ, Ehmke B, Flemmig TF. Antimicrobial effects of mechanical debridement. Periodontol 2000. 2002;28:56-71. doi: 10.1034/j.1600-0757.2002.280103.x. PMID 12013348
- [Background] Salzer S, Slot DE, Van der Weijden FA, Dorfer CE. Efficacy of inter-dental mechanical plaque control in managing gingivitis--a meta-review. J Clin Periodontol. 2015 Apr;42 Suppl 16:S92-105. doi: 10.1111/jcpe.12363. PMID 25581718
- [Background] Slot DE, Dorfer CE, Van der Weijden GA. The efficacy of interdental brushes on plaque and parameters of periodontal inflammation: a systematic review. Int J Dent Hyg. 2008 Nov;6(4):253-64. doi: 10.1111/j.1601-5037.2008.00330.x. PMID 19138177